CLINICAL TRIAL: NCT06293950
Title: Allogeneic Wharton Jelly Mesenchymal Stromal Cell (WJMSC) for Treatment of Autism
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Hanan Jafar, Principal investigator, University of Jordan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUTISM
Record Dates: First submitted 2023-05-09; First posted 2024-03-05 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Autism
Keywords: autism; WJMSC
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WJMSC (Experimental): - Patients receive three intravenous doses of MSCs (1 million/kg) every two weeks as treatment.
  Interventions: Biological: WJMSC

INTERVENTIONS:
Biological: WJMSC — - Patients receive three intravenous doses of MSCs (1 million/kg) every two weeks as treatment.

SUMMARY:
Autism spectrum disorders (ASDs) are characterized by core domains: persistent deficits in social communication and interaction; restricted, repetitive patterns of behavior, interests, or activities.

DETAILED DESCRIPTION:
Autism spectrum disorders (ASDs) are characterized by core domains: persistent deficits in social communication and interaction; restricted, repetitive patterns of behavior, interests, or activities. ASDs comprise heterogeneous and complex neuro-developmental pathologies with well-defined inflammatory conditions and immune system dysfunction. Due to neurobiological changes underlying ASD development, cell-based therapies have been proposed and applied to ASDs. Indeed, stem cells show specific immunologic properties, which make them promising candidates for ASD treatment.

ELIGIBILITY:
Inclusion Criteria:

* 14 subjects, 4-14 years of age, will be enrolled into this study, who meet the criteria for (ASD

Exclusion Criteria:

* Age > 14 years.
* Patient weighing < 10 kg.
* History of severe Allergy
* History of severe head trauma, defined by loss of consciousness or hospitalization, skull fracture, or stroke.
* Seizure within the last year before enrollment, or the need for seizure medications either at present or in the past.
* Evidence or history of severe, moderate, or uncontrolled systemic disease.
* Inability to follow the prescribed dosing and follow-up schedule.
* Use of any stimulant or non-stimulant medication or medications given for attention deficit hyperactivity disorder (ADHD) must be discontinued 7 days before the initial randomized study period.
* Subjects taking a selective serotonin reuptake inhibitor (SSRI) must be on a stable dose for a minimum of 30 days before entering the study.
* History of premature birth <35 weeks' gestation.
* Prior history of stroke in utero or other in utero insult.

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Estimated)
Dates: Start 2022-03-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
safety profile lab tests | follow-up duration is 12 months
  -patients will be monitored for any possible adverse events resulting from the injection of MSCs.

SECONDARY OUTCOMES:
efficacy change in Adult ADHD Self-Report Scale (ASRS) | follow-up duration is 12 months
  -The subjects will be monitored with ASRS at baseline, 3, 6, 9, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Abdallah Awidi, MD, Study Director — Cell Therapy Center
Locations (1):
- Cell Therapy Center, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided